CLINICAL TRIAL: NCT04602806
Title: TRACK-TBI Precision Medicine Phase 2-Option I
Brief Title: Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) Precision Medicine Phase 2 Option 1
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: W81XWH-18-2-0042
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Biomarkers; Neuroimaging; Psychological Health; Concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Psychological Well-Being; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and Serum will be collected at each of the following time points: within 6 hours of injury, and again at 12h, 24h, 2d, 3d, 5d, 2w, 6w and 3m post-injury. DNA is collected only at Day 1 of the Baseline Visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate to Severe TBI Subjects: Adult patients (age 18-65y inclusive) presenting to the Emergency Department (ED) with a history of acute TBI as per American Congress of Rehabilitation Medicine (ACRM) Criteria (i.e., patient has sustained a traumatically-induced physiological disruption of brain function).

SUMMARY:
This study is being conducted to validate early and ultra-early blood-based and novel imaging biomarkers of Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and neuroinflammation that may serve as predictive and pharmacodynamic biomarkers in a new cohort of moderate-severe TRACK-TBI subjects. The study team will enroll a cohort of moderate to severe TBI subjects (N=50), stratified according to VA/DoD criteria for these injury severities through the existing TRACK-TBI network sites to obtain novel advanced neuroimaging and more frequent biomarker sampling. Subjects will be assessed over 3 months.

DETAILED DESCRIPTION:
In 2009, the multicenter Transforming Research and Clinical Knowledge in Traumatic Brain Injury Consortium was implemented to characterize the clinical, magnetic resonance imaging (MRI), and blood-based biomarker features of TBI to inform design of next-generation precision medicine clinical trials in TBI. Over the past 10+ years, TRACK-TBI has been supported by National Institute of Neurological Disorders and Stroke (NINDS), Department of Defense (DoD), Department of Energy (DoE), the National Football League, and other philanthropic and industry partners. TRACK-TBI has enrolled >3000 control and TBI subjects across the injury spectrum at 18 US Level 1 Trauma Centers. This effort has established the world's largest collection of TBI imaging studies and bio-specimens. The study results are already being adopted into clinical research and bedside practice. The TRACK-TBI Consortium is now primed to deliver on critical military and public health knowledge gaps and needs: objective classification of TBI based on what is termed as "mechanistic" endophenotypes, e.g., diffuse axonal injury (DAI), microvascular injury (MVI), and neuroinflammation. An endophenotype is an internal phenotype discoverable by biochemical, physiological, radiological, pathological, or other techniques, which is intermediate between a complex phenotype and the presumptive genetic or environmental contribution to a disease. Endophenotypes are quantitative, continuous variables, unlike a phenotype which is usually a binary, categorical variable. These mechanistic endophenotypes, defined by imaging and blood-based biomarkers, will direct targeted treatments based on mechanism, providing the tools needed for successful execution of precision medicine clinical trials. To achieve the goal of precision medicine in TBI, it is necessary to identify subgroups of TBI patients that will respond to a targeted therapy. Investigators will assess putative blood-based and neuroimaging biomarkers for DAI, MVI, and neuroinflammation. Fluid biomarkers complement imaging markers and may provide important tools for precision medicine clinical trials. Investigators will collect acute data (early and ultra-early i.e., hours-days following injury), to validate the utility of these biomarkers in defining TBI mechanistic endophenotypes for use in clinical trials.

Specific Aim for TRACK-TBI Precision Medicine Phase 2-Option 1: To validate early and ultra-early blood based and novel imaging biomarkers of DAI, MVI, and neuroinflammation that may serve as predictive and pharmacodynamic biomarkers in a cohort of moderate-severe subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65y inclusive
* History or evidence of TBI, according to DoD-VA criteria
* Glasgow Coma Scale (GCS) 3 - 15 after resuscitation in the ED
* Head CT with evidence of trauma-related abnormality (except for isolated epidural hematoma (EDH))
* Ability to undergo MRI within 48 hours of injury
* Ability to obtain informed consent from participant or Legally Authorized Representative (LAR) within 6 hours of injury
* Fluency in English or Spanish

Exclusion Criteria:

* Unstable respiratory or hemodynamic status
* Evidence of penetrating brain injury
* Isolated EDH as only trauma-related CT abnormality
* Systemic traumatic injury that would preclude participation in study, which is expected to result in long-term disability not related to TBI
* Evidence of serious infectious complications (sepsis, bacteremia, multilobar pneumonia)
* Acute ischemic heart disease (myocardial infarction or unstable angina)
* History of syncope or hypotension
* Systolic blood pressure (SBP) < 90 mm Hg, Diastolic blood pressure (DBP)< 40 mm Hg for longer than 5 minutes
* History or evidence of active malignancy
* History of pre-existing neurologic disorder, such as dementia, mild cognitive impairment, uncontrolled epilepsy, multiple sclerosis, strokes, brain tumors, prior severe TBI, or other disorder that may confound interpretation of MRI or neuropsychological results
* History of pre-existing disabling mental illness, such as major depression or schizophrenia
* History or evidence of chronic heart failure or chronic renal failure
* Low likelihood of follow-up (e.g., participant or family indicating low interest, residence in another state or country, unhoused or lack of reliable contacts)
* Women who are pregnant or breast-feeding
* Prisoners or patients in custody
* Patients on psychiatric hold (e.g. 5150, 5250)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a population-based TBI study. All patients presenting with traumatic brain injury and receive a head CT scan as part of standard care within 6 hours of injury are initially eligible.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2030-04-09 (Estimated)

PRIMARY OUTCOMES:
Blood Specimen for Analysis of Biomarkers | < 6 hours from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | 12 hours from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | 24 hours from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | Day 2 from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | Day 3 from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | Day 5 from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | Week 4 from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | Week 6 from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
Blood Specimen for Analysis of Biomarkers | 3 Months from the time of TBI
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NfL), Tau, Interleukin 6 (IL6), Interleukin (IL10), and Tumor Necrosis Factor (TNF) will be measured to validate their utility as early predictive and pharmacodynamic biomarkers for Diffuse Axonal Injury (DAI), Microvascular Injury (MVI), and Neuroinflammation. In addition, Ubiquitin C-terminal Hydrolase L1 (UCH-L1)/Glial fibrillary acidic protein (GFAP) markers will also be assayed for comparison. All biomarkers will be measured in picograms/milliliter (pg/mL).
3 Tesla Brain Structural and Functional Magnetic Resonance Imaging (MRI) | Within 24-48 hours from the time of TBI
  This study aims to validate early and ultra-early novel imaging biomarkers in the acute phase after injury. In addition to volumetrics, Diffuse Tensor Imaging (DTI) and Resting State Functional Magnetic Resonance Imaging (rs-fMRI), the MRI protocol will incorporate novel imaging measures of axonal density using neurite density index (NDI) from Neurite Orientation Dispersion And Density Imaging (NODDI) analysis of multi-shell diffusion MRI, cerebral blood flow using Arterial Spin Labeled (ASL) perfusion, and neuroinflammation using free water content isotropic diffusion fraction (FISO) from NODDI analysis of multi-shell diffusion MRI.
3 Tesla Brain Structural and Functional Magnetic Resonance Imaging (MRI) | 2 Weeks from the time of TBI
  This study aims to validate early and ultra-early novel imaging biomarkers in the acute phase after injury. In addition to volumetrics, Diffuse Tensor Imaging (DTI) and Resting State Functional Magnetic Resonance Imaging (rs-fMRI), the MRI protocol will incorporate novel imaging measures of axonal density using neurite density index (NDI) from Neurite Orientation Dispersion And Density Imaging (NODDI) analysis of multi-shell diffusion MRI, cerebral blood flow using Arterial Spin Labeled (ASL) perfusion, and neuroinflammation using free water content isotropic diffusion fraction (FISO) from NODDI analysis of multi-shell diffusion MRI.
3 Tesla Brain Structural and Functional Magnetic Resonance Imaging (MRI) | 3 Months from the time of TBI
  This study aims to validate early and ultra-early novel imaging biomarkers in the acute phase after injury. In addition to volumetrics, Diffuse Tensor Imaging (DTI) and Resting State Functional Magnetic Resonance Imaging (rs-fMRI), the MRI protocol will incorporate novel imaging measures of axonal density using neurite density index (NDI) from Neurite Orientation Dispersion And Density Imaging (NODDI) analysis of multi-shell diffusion MRI, cerebral blood flow using Arterial Spin Labeled (ASL) perfusion, and neuroinflammation using free water content isotropic diffusion fraction (FISO) from NODDI analysis of multi-shell diffusion MRI.

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | 2 Weeks from the time of TBI
  The GOSE provides an overall measure of functional status based on information on cognition, independence, employability, and social/community participation collected via structured interview. Individuals are described by one of the eight outcome categories: Dead (1); Vegetative State (2); Lower Severe Disability (3); Upper Severe Disability (4); Lower Moderate Disability (5); Upper Moderate Disability (6); Lower Good Recovery (7) and Upper Good Recovery (8). Good Recovery is defined as a score of 7-8, Moderate Disability is defined by a score of 5-6 and Severe Disability is defined by a score of 3-4.
Glasgow Outcome Scale Extended (GOSE) | 6 Weeks from the time of TBI
  The GOSE provides an overall measure of functional status based on information on cognition, independence, employability, and social/community participation collected via structured interview. Individuals are described by one of the eight outcome categories: Dead (1); Vegetative State (2); Lower Severe Disability (3); Upper Severe Disability (4); Lower Moderate Disability (5); Upper Moderate Disability (6); Lower Good Recovery (7) and Upper Good Recovery (8). Good Recovery is defined as a score of 7-8, Moderate Disability is defined by a score of 5-6 and Severe Disability is defined by a score of 3-4.
Glasgow Outcome Scale Extended (GOSE) | 3 Months from the time of TBI
  The GOSE provides an overall measure of functional status based on information on cognition, independence, employability, and social/community participation collected via structured interview. Individuals are described by one of the eight outcome categories: Dead (1); Vegetative State (2); Lower Severe Disability (3); Upper Severe Disability (4); Lower Moderate Disability (5); Upper Moderate Disability (6); Lower Good Recovery (7) and Upper Good Recovery (8). Good Recovery is defined as a score of 7-8, Moderate Disability is defined by a score of 5-6 and Severe Disability is defined by a score of 3-4.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey T Manley, MD, PhD, Study Director — University of California, San Francisco; Claudia S Robertson, MD, Study Director — Baylor College of Medicine; David O Okonkwo, MD, PhD, Study Director — University of Pittsburgh Medical Center; Ramon Diaz-Arrastia, MD, PhD, Study Director — University of Pennsylvania; Nancy R Temkin, PhD, Study Director — University of Washington; Pratik Mukherjee, MD, PhD, Study Director — University of California, San Francisco; Joseph T Giacino, PhD, Study Director — Harvard Medical School, Spaulding Rehabilitation Hospital; Murray B Stein, MD, MPH, Study Director — University of California, San Diego; Mike McCrea, PhD, ABPP, Principal Investigator — Medical College of Wisconsin; Ramesh Grandhi, MD, MS, Principal Investigator — University of Utah
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - University of Pennsylvania/Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
* The TRACK TBI investigators have created a Data Use Agreement/Human Materials Transfer Agreement (DUA/HTMA) for TRACK-TBI Research Collaborations. This Agreement is for the use of clinical data, neuroimaging, and bio-specimens collected by the TRACK-TBI investigators. All Research Collaborators can submit a written request to the TRACK-TBI Executive Committee.
  * This study involves research in the area of traumatic brain injury (TBI). The Department of Defense, in collaboration with the National Institutes of Health, has developed the Federal Interagency Traumatic Brain Injury Research (FITBIR) Informatics System, a central repository and resource for sharing data to promote collaboration, accelerate research, and advance knowledge on the characterization, prevention, diagnosis, and treatment of TBI. The TRACK-TBI Investigators will share study data via FITBIR in accordance with FITBIR policy and procedures.
Time Frame: Data will become available after study completion.
Access Criteria: * All Research Collaborations with TRACK-TBI begins with a written request submitted to the TRACK-TBI Executive Committee. The Research Collaboration Proposal form is attached as Appendix 1 in the Research Collaboration Policy available on the TRACK-TBI website.
  * Access to FITBIR data will be according to FITBIR policies found at https://fitbir.nih.gov/jsp/about/policy.jsp
URL: https://tracktbi.ucsf.edu/collaboration-opportunities

REFERENCES:
- [Background] Maas AI, Roozenbeek B, Manley GT. Clinical trials in traumatic brain injury: past experience and current developments. Neurotherapeutics. 2010 Jan;7(1):115-26. doi: 10.1016/j.nurt.2009.10.022. PMID 20129503
- [Background] Teasdale G, Jennett B. Assessment and prognosis of coma after head injury. Acta Neurochir (Wien). 1976;34(1-4):45-55. doi: 10.1007/BF01405862. PMID 961490
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Background] Maas AI, Harrison-Felix CL, Menon D, Adelson PD, Balkin T, Bullock R, Engel DC, Gordon W, Orman JL, Lew HL, Robertson C, Temkin N, Valadka A, Verfaellie M, Wainwright M, Wright DW, Schwab K. Common data elements for traumatic brain injury: recommendations from the interagency working group on demographics and clinical assessment. Arch Phys Med Rehabil. 2010 Nov;91(11):1641-9. doi: 10.1016/j.apmr.2010.07.232. PMID 21044707
- [Background] Manley GT, Diaz-Arrastia R, Brophy M, Engel D, Goodman C, Gwinn K, Veenstra TD, Ling G, Ottens AK, Tortella F, Hayes RL. Common data elements for traumatic brain injury: recommendations from the biospecimens and biomarkers working group. Arch Phys Med Rehabil. 2010 Nov;91(11):1667-72. doi: 10.1016/j.apmr.2010.05.018. PMID 21044710
- [Background] Duhaime AC, Gean AD, Haacke EM, Hicks R, Wintermark M, Mukherjee P, Brody D, Latour L, Riedy G; Common Data Elements Neuroimaging Working Group Members, Pediatric Working Group Members. Common data elements in radiologic imaging of traumatic brain injury. Arch Phys Med Rehabil. 2010 Nov;91(11):1661-6. doi: 10.1016/j.apmr.2010.07.238. PMID 21044709
- [Background] Whyte J, Vasterling J, Manley GT. Common data elements for research on traumatic brain injury and psychological health: current status and future development. Arch Phys Med Rehabil. 2010 Nov;91(11):1692-6. doi: 10.1016/j.apmr.2010.06.031. PMID 21044713
- [Background] Almasy L, Blangero J. Endophenotypes as quantitative risk factors for psychiatric disease: rationale and study design. Am J Med Genet. 2001 Jan 8;105(1):42-4. PMID 11424994
- [Background] O'Neil ME, Carlson KF, Storzbach D, Brenner LA, Freeman M, Quinones AR, Motu'apuaka M, Kansagara D. Factors associated with mild traumatic brain injury in veterans and military personnel: a systematic review. J Int Neuropsychol Soc. 2014 Mar;20(3):249-61. doi: 10.1017/S1355617714000204. PMID 24622505
- [Background] Alsop DC, Detre JA, Golay X, Gunther M, Hendrikse J, Hernandez-Garcia L, Lu H, MacIntosh BJ, Parkes LM, Smits M, van Osch MJ, Wang DJ, Wong EC, Zaharchuk G. Recommended implementation of arterial spin-labeled perfusion MRI for clinical applications: A consensus of the ISMRM perfusion study group and the European consortium for ASL in dementia. Magn Reson Med. 2015 Jan;73(1):102-16. doi: 10.1002/mrm.25197. Epub 2014 Apr 8. PMID 24715426
- [Background] Dikmen S, Machamer J, Miller B, Doctor J, Temkin N. Functional status examination: a new instrument for assessing outcome in traumatic brain injury. J Neurotrauma. 2001 Feb;18(2):127-40. doi: 10.1089/08977150150502578. PMID 11229707
- [Background] McCrea M, Kelly JP, Randolph C. Standardized Assessment of Concussion (SAC): Manual for Administration, Scoring and Interpretation. 2nd ed. Waukesha, WI: CNS Inc; 2000. [Google Scholar]
- [Background] Smith GP, Burger GK. Detection of malingering: validation of the Structured Inventory of Malingered Symptomatology (SIMS). J Am Acad Psychiatry Law. 1997;25(2):183-9. PMID 9213290
- [Background] Reitan, R.M. and D. Wolfson, The Halstead-Reitan neuropsychological test battery: Theory and clinical interpretation. Vol. 4. 1985: Reitan Neuropsychology.
- [Background] Finkelstein E, Corso P, Miller T and Associates. The Incidence and Economic Burden of Injuries in the United States. New York (NY): Oxford University Press; 2006.
- See also: Access to FITBIR data will be according to FITBIR policies. — https://fitbir.nih.gov/content/access-data